CLINICAL TRIAL: NCT06230822
Title: A Phase I Open Label, Dose Escalation Study to Characterize the Safety, Tolerability, and Efficacy of VUM02 Injection in Subjects With Idiopathic Pulmonary Fibrosis
Brief Title: Safety, Tolerability and Efficacy of VUM02 Injection in Treatment of Idiopathic Pulmonary Fibrosis (IPF)
Acronym: DEVIF-I
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wuhan Optics Valley Vcanbiopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Vcanbio Cell and Gene Engineering Corp., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VUM02-IPF-01
Record Dates: First submitted 2023-12-29; First posted 2024-01-30 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: VUM02 Injection (hUCT-MSCs)+Conventional treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VUM02 Injection (hUCT-MSCs)+Conventional treatment (Experimental): 3 predefined dose groups: 5x10^7 cells/person/time, 1x10^8 cells/person/time and 2x10^8 cells/person/time, administered intravenously on D0, D3 and D6 for a total of 3 doses.
  Interventions: Drug: VUM02 Injection

INTERVENTIONS:
Drug: VUM02 Injection — VUM02 Injection will be administered intravenously every 3 days for a total of 3 doses.
  Other Names: Human Umbilical Cord Tissue-derived Mesenchymal Stem Cells Injection

SUMMARY:
This study is a single-arm, multiple-dose, dose-escalation, open-label multicenter clinical trial, aiming to evaluate the safety, tolerability, and preliminary efficacy of VUM02 Injection for treatment of idiopathic pulmonary fibrosis (IPF). VUM02 Injection (Human Umbilical Cord Tissue-derived Mesenchymal Stem Cells Injection, hUCT-MSC) is an allogeneic cell therapy product comprising culture-expanded Mesenchymal Stem Cells derived from the human umbilical cord tissue. The product is cryopreserved with the amount of 5 x 10^7 cells per 10 mL per bag (5 x 10^6 cells/mL). This study is a multiple-dose tolerability study following the "3+3" dose escalation principle and progressing from the low-dose group to the high-dose group sequentially. Three to six patients will be enrolled in each dose group and administered every 3 days for a total of 3 doses.

DETAILED DESCRIPTION:
This trial includes three predefined dose groups: low dose (5E7 cells/person/time), medium dose (1E8 cells/person/time), and high dose (2E8 cells/person/time) groups, for a multiple-dose tolerability study. Each dose group undergoes an initial safety and tolerability assessment with a single dose. After receiving the initial dose, subjects undergo safety evaluations on Day 3 (including symptom assessment, physical examination, vital signs monitoring, 12-lead electrocardiogram, hematology, urinalysis, blood biochemistry, and coagulation function tests). The decision to proceed with subsequent administrations for subjects who have received the initial dose is made through discussion between the investigator and the sponsor (and/or CRO medical staff) based on safety profiles.

This study follows the "3+3" dose escalation principle, progressing from the low-dose group to the high-dose group sequentially. The sample size may be adjusted based on the actual circumstances of the trial, with each subject receiving only one corresponding dose. During the study, a Safety Monitoring Committee (SMC) will be established, consisting of the investigators and representatives from the sponsor. The SMC will review the safety data generated during the study and make decisions regarding dose escalation, modification of escalation doses, alteration of dosing regimens, or study discontinuation. Only after all subjects in the preceding dose group have completed the dose-limiting toxicity (DLT) observation, and the SMC confirms that the dose escalation criteria are met, the enrollment for the next dose group will begin.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for this trial:

1. Gender unrestricted, aged between 40 and 75 years old (inclusive);
2. Diagnosed with IPF according to the 2022 Idiopathic Pulmonary Fibrosis (an Update) and Progressive Pulmonary Fibrosis in Adults: An Official ATS/ERS/JRS/ALAT Clinical Practice Guideline.
3. In the 3 months prior to administration, determined by the investigator to have stable disease, with diffusing capacity of the lung for carbon monoxide (DLCO) between 30% and 79% of the predicted value (adjusted for Hb), FVC/predicted ≥50%, and forced expiratory volume in one second (FEV1)/FVC ≥0.70;
4. Allowed to enroll are the patients who have been treated according to the current standard treatment plan for IPF and have maintained the treatment for at least 3 months;
5. Good compliance, able to understand and cooperate with pulmonary function test procedures, willing to participate voluntarily in the trial according to the protocol requirements, and understand and sign the informed consent form voluntarily.

Exclusion Criteria:

Patients meeting any of the following criteria are not eligible for this trial:

1. Allergic to any ingredient of the product;
2. Suffering from interstitial lung diseases (ILD) other than IPF, including but not limited to: any other type of interstitial pneumonia; lung diseases related to exposure to fibrogenic agents or other environmental toxins or drugs (such as amiodarone, bleomycin, or methotrexate); other types of occupational lung diseases; granulomatous lung diseases; systemic diseases including vasculitis, infectious diseases (i.e., tuberculosis), and connective tissue diseases, or a history of prior pulmonary resection;
3. During the screening period, having any of the following pulmonary diseases: asthma, pulmonary embolism, pneumothorax; lung cancer, obstructive bronchitis, or other active lung diseases; a known history of immune system diseases (such as thymic diseases, systemic lupus erythematosus); acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
4. Chest HRCT during the screening period shows emphysema area > fibrosis area;
5. Previously received stem cell therapy or intolerant to cell therapy;
6. Received unstable standard of care for IPF within the 3 months prior to screening;
7. Used non-biological drugs with cell proliferation inhibition or immunosuppressive/immunomodulatory effects during the 3 months prior to screening, such as Mycophenolate Mofetil, cyclophosphamide, tacrolimus, and JAK inhibitors, as well as other Chinese herbal medicines with immunomodulatory effects;
8. Used biologics such as rituximab, TNF-α monoclonal antibodies, and IFN-γ monoclonal antibodies within the 6 months prior to screening;
9. Used anticoagulant drugs, sildenafil, bosentan, macitentan, imatinib, and other drugs for treating IPF within the 4 weeks prior to screening;
10. Participated in interventional clinical studies within the 3 months or within the half-life of 5 drugs (whichever is longer) before screening;
11. Hospitalized 2 or more times in the past year due to acute exacerbation of IPF;
12. Had a lung infection within the past month;
13. Had a history of invasive or non-invasive mechanical ventilation, or currently require oxygen therapy (oxygen therapy time >15 h/d);
14. Smoked within the past 3 months or cannot quit smoking during the trial;
15. The expected survival period may be less than 1 year judged by investigator;
16. Laboratory tests meet any of the following criteria: white blood cell count less than 3.5×109/L or neutrophils less than 1.5×109/L for any reason; hemoglobin (HGB) ≤90 g/L; fibrinogen (FIB) ≤0.5×LLN; alanine aminotransferase (ALT) >2×ULN, aspartate aminotransferase (AST) >2×ULN, total bilirubin (TBIL) >1.5×ULN, direct bilirubin (DBIL) >1.5×ULN, blood creatinine (Cr) >1.5×ULN;
17. Evidence suggests that the subject currently has digestive system, urinary system, cardiovascular system, hematological system, nervous system, psychiatric, or metabolic diseases that may affect safety, such as severe kidney disease requiring blood dialysis or peritoneal dialysis; advanced hepatitis or cirrhosis; severe heart failure (NYHA Grade III and IV); poorly controlled hypertension (≥180/100 mmHg); severe pulmonary heart disease or pulmonary arterial hypertension considered by the investigators to affect the evaluation of the trial results;
18. Have various malignant tumors or a history of malignant tumors;
19. 12-lead electrocardiogram shows severe arrhythmias (such as ventricular tachycardia, frequent supraventricular tachycardia, atrial fibrillation, and atrial flutter) or degree II and above atrioventricular block;
20. Positive results in serological tests (HBsAg, HCV antibodies, HIV antibodies, syphilis spirochete antibodies), among which carriers of hepatitis B virus, stable patients with hepatitis B (DNA titer ≤2000 IU/mL or copy number <1000 copies/mL) after drug treatment, and cured patients with hepatitis C (negative HCV RNA) can be enrolled after being judged eligible by the investigator;
21. Pregnant or lactating women, or those with a positive result in the screening period for beta-human chorionic gonadotropin (β-HCG) testing; or male subjects of childbearing potential and female subjects of childbearing age who are unable and unwilling to take effective non-drug contraceptive measures during the study and 6 months after the end of the study;
22. Subjects deemed inappropriate for entry into this study by the investigator.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of cell therapy-related adverse events (AEs) as assessed by CTCAE (V5.0) | 28 days
  Incidence and severity of cell therapy-related adverse events (AEs) from the first dosing to 28 days after the last dosing
Maximum tolerated dose (MTD) | 28 days
  Maximum tolerated dose (MTD) with multiple administrations.

SECONDARY OUTCOMES:
Incidence and severity of treatment- emergent adverse events | 24 weeks
  Incidence and severity of cell treatment-emergent adverse events (AEs) as assessed by CTCAE v5.0 from the first dosing to 24 weeks after the last dosing.
DLCO changes from baseline | At baseline, 1, 4, 12 and 24 weeks
  Changes from baseline in the percentage of diffusing capacity of the lung for carbon monoxide (DLCO) to the predicted value at 1 week, 4 weeks, 12 weeks, and 24 weeks after the last dosing.
FVC changes from baseline | At baseline, 1, 4, 12 and 24 weeks
  Changes from baseline in the forced vital capacity (FVC) at 1 week, 4 weeks, 12 weeks, and 24 weeks after the last dosing.
Exercise capacity changes from baseline | At baseline, 1, 4, 12 and 24 weeks
  Changes from baseline in the 6-minute walk test distance at 1 week, 4 weeks, 12 weeks, and 24 weeks after the last dosing.
St. George's Respiratory Questionnaire | At baseline, 1, 4, 12 and 24 weeks
  Changes from baseline in the St. George's Respiratory Questionnaire (SGRQ) total score at 1 week, 4 weeks, 12 weeks, and 24 weeks after the last dosing. The SGRQ is a 50-item questionnaire developed to measure health status (quality of life). Scores are calculated for three domains: Symptoms, Activity and Impacts. The total score (summed weights) can range from 0 to 100 with a lower score denoting a better health status.
Symptoms of dyspnea | At baseline, 1, 4, 12 and 24 weeks
  Changes from baseline in the dyspnea score at 1 week, 4 weeks, 12 weeks, and 24 weeks after the last dosing.
Symptoms of cough | At baseline, 1, 4, 12 and 24 weeks
  Changes from baseline in the cough score at 1 week, 4 weeks, 12 weeks, and 24 weeks after the last dosing.
Tumor biomarkers | At baseline, 12 and 24 weeks
  Changes from baseline in the lung tumor markers of CYFRA21-1, NSE, SCC, CEA and CA125 at 12 weeks and 24 weeks after the last dosing.
Chest imaging changes | At baseline, 12 and 24 weeks
  Changes from baseline in the chest HRCT score at 12 weeks and 24 weeks after the last dosing.
Acute exacerbations of IPF | 24 weeks
  Frequency and severity of acute exacerbations of IPF from the first dosing to 24 weeks after the last dosing.
T lymphocyte subpopulations | At baseline, 1, 4 and 12 weeks
  Changes from baseline in the percentages of CD3+, CD4+, CD8+, CD4+/CD8+ in peripheral blood at 1 week, 4 weeks, and 12 weeks after the last dosing.
IgG and IgM levels | At baseline, 12 or 4 weeks
  Changes from baseline in IgG levels in peripheral blood up to 12 weeks after the last dosing; Changes from baseline in IgM levels in peripheral blood up to 4 weeks after the last dosing.
Inflammatory cytokines | At baseline, 1, 4 and 12 weeks
  Changes from baseline in the cytokines of TNF-α, IFN-γ, TGF-β, IL-1, IL-2, IL-4, IL-5, IL-6 and CCL2 in peripheral blood at 1 week, 4 weeks, and 12 weeks after the last dosing.
Serum complement levels | At baseline, 1, 4 and 12 weeks
  Changes from baseline in the serum complements of C3 and C4 in peripheral blood at 1 week, 4 weeks, and 12 weeks after the last dosing.
Blood proteomics analysis | At baseline, 1, 4, 12 and 24 weeks
  Changes from baseline in the blood proteomic analysis at 1 week, 4 weeks, 12 weeks, and 24 weeks after the last dosing.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Peking University Third Hospital, Beijing
  - West China Hospital of Sichuan University, Chengdu
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The First People's Hospital of Kashi Prefecture, Xinjiang, Kashgar